CLINICAL TRIAL: NCT01097135
Title: Prospective, Randomized Clinical Study to Evaluate the Efficacy of 2 Surgical Skin Preparations in Reducing Wound Drainage Following Total Joint Arthroplasty
Brief Title: Evaluating the Effectiveness of 2 Surgical Skin Preparation Methods in Reducing Surgical Wound Drainage After Total Hip or Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, Tiffany Morrison, MS, Manager, Clinical Trials, Rothman Institute, Rothman Institute Orthopaedics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIFJPAR-10-02
Record Dates: First submitted 2010-03-30; First posted 2010-04-01 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Drainage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Standard surgical skin preparation (No Intervention)
- Standard Surgical Skin Preparation with Duraprep (Active Comparator): standard surgical skin prep
  Interventions: Drug: Duraprep Surgical Solution

INTERVENTIONS:
Drug: Duraprep Surgical Solution
  Arms: Standard Surgical Skin Preparation with Duraprep

SUMMARY:
Surgical skin complications can be costly and could contribute to extended in-patient stay following total joint replacement or even the need for re-admission. If efficacy in reducing the incidence of post-operative wound drainage and, in turn, surgical wound complications can be demonstrated, it may also reduce the length of hospital stay and the need for revision surgery or readmission. The aim of this research is to investigate the incidence of post-operative wound drainage following elective total joint arthroplasty using two surgical skin preparation protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able and willing to provide informed consent
2. Male and non-pregnant, non-lactating, postmenopausal or surgically sterilized female subjects between the ages of 18-80 years old.
3. Subjects deemed able to comply with study visit schedule and procedures.
4. Subjects undergoing elective total hip arthroplasty or elective total knee arthroplasty.

Exclusion Criteria:

1. Subjects undergoing revision, unicompartmental, bilateral total knee arthroplasty or bilateral total hip arthroplasty.
2. Subjects undergoing non-elective total joint procedures.
3. Pregnant, lactating females, or females of childbearing potential not willing to practice an effective method of contraception.
4. Subjects with known allergies or previous skin reaction to iodine povacrylex

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the rate of wound drainage following total joint arthroplasty (TJA) until discharge in both treatment groups | Up to one year following surgery
  Starting on post operative day 1 (the first day following surgery), at the time of the surgical dressings are removed and changed, assessments will be made to determine level of post-operative wound drainage following TJA.

SECONDARY OUTCOMES:
The secondary objectives will focus on wound assessment and signs and symptoms of infection from TJA until discharge. | until hospital discharge
Length of hospital stay | until hospital discharge
Need for readmission or reoperation for up to 6 weeks following TJA | 6 weeks post-op
Incidence of surgical skin infection at the first post-operative visit (6 weeks following surgery) | 6 weeks post-op
Incidence of skin blistering. | up to one year post-op
Scar cosmesis at the first post-operative visit. | up to 6 weeks post-op

CONTACTS AND LOCATIONS:
Overall Officials: Javad Parvizi, MD, FRCS, Principal Investigator — Rothman Institute
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States